CLINICAL TRIAL: NCT04795817
Title: A Prospective Single Center Investigation of the da Vinci® SP™ Surgical System for Transoral Robotic Surgery (TORS) for Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: Treatment of Obstructive Sleep Apnea (OSA) With the da Vinci® SP™ Surgical System
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: dV SP-TORS OSA
Record Dates: First submitted 2021-02-01; First posted 2021-03-12 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Single arm: Subjects will undergo TORS benign base of tongue resection procedures (i.e., partial glossectomy, epiglottoplasty, epiglottectomy, and/or lingual tonsillectomy) for the treatment of OSA
  Interventions: Device: Transoral Robotic Surgery

INTERVENTIONS:
Device: Transoral Robotic Surgery — Subjects will undergo TORS benign base of tongue resection procedures (i.e., partial glossectomy, epiglottoplasty, epiglottectomy, and/or lingual tonsillectomy) for the treatment of OSA. Concomitant non-robotic surgical procedures may also be performed as part of the subject's treatment for OSA, and can include one or more of the following: uvulopalatopharyngoplasty (UPPP), lateral pharyngoplasty, expansion sphincter pharyngoplasty, palatine tonsillectomy, or a modified uvulopalatoplasty. Nasal surgery such as septoplasty or turbinoplasty can be combined if it is needed.

SUMMARY:
It is a prospective, single center, single-arm clinical study to enroll a maximum of 25 subjects.

DETAILED DESCRIPTION:
It is a prospective, single center, single-arm clinical study to enroll a maximum of 25 subjects. The objective of this study is to evaluate the clinical utility of the da Vinci® SP™ Surgical System, instruments and accessories in TORS benign base of tongue resection procedures for the treatment of moderate to severe OSA. da Vinci® SP™ Surgical System, instruments and accessories are the approved medical device product by MFDS (Ministry of Food and Drug Safety, Republic of Korea).

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 80 years old
* Subject with BMI ≤ 35
* Subject with moderate to severe sleep apnea, defined as 15 or more AHI events/hour
* Subject who has failed or is unable to tolerate CPAP therapy
* Subject diagnosed with OSA due to redundant base of tongue tissue
* Subject must be a suitable candidate for base of tongue resection surgery
* Subject who is willing and able to provide written informed consent
* Subject who is willing and able to comply with the study protocol requirements

Exclusion Criteria:

* Subject with a poor mouth opening or trismus
* Subject with evidence of any primary cancers or metastatic disease, other than skin cancers
* Subject who has had a surgical resection and/or chemoradiation therapy for oropharyngeal cancer
* Subject with congenital malformations in the larynx, throat or tongue
* Subject with an American Society of Anesthesiologists (ASA) score of Grade 4 or above during preoperative evaluation
* Subject for whom any additional surgeries are planned for OSA within the study period, after the surgery in which the da Vinci SP System was used
* Subject who is mentally handicapped or with a psychological disorder or severe systemic illness, that would preclude compliance with study requirements or ability to provide informed consent
* Subject is pregnant or suspected to be pregnant

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Subject who has failed or is unable to tolerate CPAP therapy
  * Subject who is diagnosed with OSA due to redundant base of tongue tissue
  * Subject who has moderate to severe sleep apnea, defined as 15 or more AHI events/hour
  * Subject who has planned a tongue base resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Type 1 Polysomnography (PSG) | Pre-operative (within 12 months prior to surgery)
  Type I PSG measurements demonstrating Apnea Hypopnea Index (AHI) reduction.
Type 1 Polysomnography (PSG) | 90-150 days after surgery
  Type I PSG measurements demonstrating Apnea Hypopnea Index (AHI) reduction.

SECONDARY OUTCOMES:
Total operative time | Intra-Operative Assessment
  defined as the time the patient spends in the operating room (OR), i.e. OR "In and Out" time. This includes the patient prep time, anesthesia time, robotic docking time, robotic procedure time and time taken for non-robotic concomitant procedures, which are part of the multi-level surgical treatment approach for that particular patient.
Robotic procedure time | Intra-Operative Assessment
  defined as time from docking the robot at the initiation of surgery to undocking at the completion of surgery.
Estimated blood loss (EBL) | Intra-Operative Assessment
  defined as the estimated amount of blood loss
Postoperative hemorrhage | Intra-Operative Assessment
  categorized using the Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Blood transfusions | Intra-Operative Assessment
  defined as whether a blood transfusion was applied or not.
Length of hospital stay (LOS) | Admission to the hospital to discharge from the hospital (check out time), up to an approximate of one week
  Duration of hospital say(from admission to discharge)
Volume of resected tissue | Immediately after surgery
  measured using the volume displacement method
Conversion rate | Intra-Operative Assessment
  from da Vinci SP surgery to any alternate method required to complete the indicated procedure.
Change in Apnea index (AI) | Pre-operative Assessments & Post-Operative (3 months +60 days) Assessment
  at 3 months (+60 days) post-surgery compared to baseline
Change in Hypopnea index (HI) | Pre-operative Assessments & Post-Operative (3 months +60 days) Assessment
  at 3 months (+60 days) post-surgery compared to baseline
Change in Percentages of sleep stages (N1, N2, N3, R) | Pre-operative Assessments & Post-Operative (3 months +60 days) Assessment
  at 3 months (+60 days) post-surgery compared to baseline
Change in Lowest oxygen saturation (LSAT) | Pre-operative Assessments & Post-Operative (3 months +60 days) Assessment
  at 3 months (+60 days) post-surgery compared to baseline
Change in Percent sleep time below 90 percent oxygen saturation (ST90) | Pre-operative Assessments & Post-Operative (3 months +60 days) Assessment
  at 3 months (+60 days) post-surgery compared to baseline
Change in Epworth Sleepiness Scale (ESS) | Pre-operative Assessments & Post-Operative (3 months +60 days) Assessment
  at 3 months (+60 days) post-surgery compared to baseline
Change in Stanford Sleepiness Scale (SSS) | Pre-operative Assessments & Post-Operative (3 months, +60 days) Assessment
  at 3 months (+60 days) post-surgery compared to baseline
Change in Berlin Questionnaire | Pre-operative Assessments & Post-Operative (3 months, +60 days) Assessment
  at 3 months (+60days) compared to baseline
Change in MDADI (MD Anderson Dysphagia Inventory) | Pre-operative Assessments & Post-Operative (3 months, +60 days) Assessment
  at 3 months (+60days) compared to baseline
Adverse Events (AE) | Through study conclusion (3 month follow up +60 days)
  Assessment of all reported adverse events (AE) within 3 months +60 days (90-150 days) post-surgery. Summarizing the incidence and frequency of all reported adverse events and categorizing them using CTCAE v4.03
Change in Upper airway volume | Pre-operative Assessment, Post-operative (within 30days ±14 days from surgery) Assessment & Post-Operative (3 months, +60 days) Assessment
  measured by CT scan as optional

CONTACTS AND LOCATIONS:
Overall Officials: HyungJu Cho, M.D., Ph.D., Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jeong Y, Rha MS, Kim CH, Cho HJ. First Prospective Study on Single-Port Robotic Tongue Base Resection for Sleep Apnea. Head Neck. 2025 Apr;47(4):1071-1078. doi: 10.1002/hed.28007. Epub 2024 Nov 22. PMID 39576059